CLINICAL TRIAL: NCT04583800
Title: Prediction of Heart Failure and Cognitive Decline in Type 2 Diabetes : Longitudinal Cohort Study of Immuno-inflammation, Cardiac Energetics and Cognition.PreciDIAB-HEART&BRAIN
Brief Title: Prediction of Heart Failure and Cognitive Decline in Type 2 Diabetes
Acronym: PreciDIAB-H&B
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_66; 2020-A01452-37 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure; Cognitive Decline
Keywords: Dementia; Stroke Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type 2 diabetes is a risk factor of heart failure and cognitive decline. Heart failure at its early stage is often silent. At present, primary prevention for heart failure is not available. Our aim is to identify diabetic patients at risk of heart failure in order to develop personalized preventive strategies.

Type 2 diabetes is vascular and metabolic risk factor for cognitive decline though a direct lesional effect but also through an interaction with underlying neurodegenerative lesions. Our aim is to identify diabetic patients at risk of cognitive decline in order to develop personalized preventive strategies

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Persons able to understand and object to the information provided.
* Type 2 diabetic patient free of heart failure ≥stade B
* Patient affiliated with a social security scheme.
* Patient agreeing to sign the informed consent form

Exclusion Criteria:

* Patient with dementia
* Patient with at least one of the criteria for heart failure ≥stade B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 2 diabetes and free of heart failure (≥stade B).
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Heart failure (≥ stade B). | at 48 months

SECONDARY OUTCOMES:
Cognitive decline (composite endpoint) | at 48 months
  * a decrease in cognitive performance quantified at 1.5 standard deviation on at least 1 neuropsychological test within a cognitive domain (attention and speed of information processing, memory, executive functions) compared to the neuropsychological assessment performed at inclusion.
  * Appearance of dementia defined as a cognitive disorder highlighted in the neuropsychological evaluation carried out at the end of the study leading to a loss of functional autonomy in activities of daily living defined by the loss of at least 1 point on the activities of daily living ADL scale (DSM V).
Major cardio-neuro-vascular events | at 48 months
  cardioneurovascular event (composite endpoint) defined by the occurrence of death from any cause, myocardial infarction, stroke (ischemic or hemorrhagic), acute limb ischemia or a doubling of creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Cordonnier, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France